CLINICAL TRIAL: NCT00384046
Title: 24-Week Study to Evaluate the Efficacy/Safety of Transdermal Testosterone in Naturally Menopausal Women With Hypoactive Sexual Desire Disorder Receiving Systemic Transdermal Estrogen Therapy.
Brief Title: Testosterone Therapy in Naturally Menopausal Women With Low Sexual Desire Receiving Transdermal Estrogen
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Warner Chilcott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2005108
Record Dates: First submitted 2006-10-03; First posted 2006-10-04 (Estimated); Last update posted 2013-04-17 (Estimated); Status verified 2013-04

CONDITIONS: Hypoactive Sexual Desire Disorder
MeSH Terms: conditions — Sexual Dysfunctions, Psychological | interventions — Testosterone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 300mcg/day testosterone
  Interventions: Drug: Testosterone
- 2 (Placebo Comparator): Placebo arm
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Testosterone — patch, 300 mcg/day testosterone, patch changed every 3-4 days, 24 weeks
  Arms: 1
Drug: Placebo — patch, placebo, patch changed every 3-4 days, 24 weeks
  Arms: 2

SUMMARY:
The purpose of this study is to examine whether the transdermal testosterone system (TTS) is effective and safe in the treatment of hypoactive sexual desire disorder (HSDD) in postmenopausal women who are on transdermal estrogen.

DETAILED DESCRIPTION:
This is a randomised, double-blind, placebo-controlled, parallel-group, multicentre, 24 week study to be conducted in approximately 300 patients at approximately 14 clinical sites in the UK, 6 sites in Australia, 5 sites in Germany, and 2 sites in Canada. Women will be randomised 1:1 to receive 300 mcg/day TTS or placebo for a 24 week period. Consistent with previous phase III studies, efficacy will be assessed over 24 weeks using the Sexual Activity Log (SAL), and at 12 and 24 weeks using the Profile of Female Sexual Function (PFSF) and Personal Distress Scale (PDS). Safety will be assessed over the entire 24 weeks. Hormone data (free and total testosterone, total estradiol, and sex hormone binding globulin) will be collected at Weeks -4 and 24. The total duration of treatment for each patient is 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Women will be screened for study participation according to the following inclusion criteria at Week -4. Eligible women must be a woman one year post menopausal, 40-70 years old in general good health on transdermal HRT and in a stable monogamous sexual relationship with low sexual desire causing distress.

Exclusion Criteria:

* Women will be screened for study participation according to the following exclusion criteria at Week -4 or as specified. Eligible women must not have any medical, physical, psychological, or pharmacological condition that could confound safety or efficacy.

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2006-11; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
To assess the efficacy of the TTS by measuring change in frequency of total satisfying episodes. The safety assessment of TTS with various parameters. | Assessment at 12 and 24 weeks

SECONDARY OUTCOMES:
To assess the efficacy of the TTS as measured by the following parameters: changes in sexual desire, personal distress, and other domains of PFSF and SAL questionnaires. | Assessment at 12 and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Imran A Lodhi, MD, Study Director — Procter and Gamble
Locations (25):
- Australia (6):
  - Research Facility, Ashfield, New South Wales
  - Research Facility, Gordon, New South Wales
  - Research Facility, Randwick, New South Wales
  - Research Facility, Dulwich, South Australia
  - Research Facility, Prahran, Victoria
  - Research Facility, Nedlands, Western Australia
- Research Facility, Freiburg, DEU, Botswana
- Canada (2):
  - Research Facility, Montreal, Quebec
  - Research Facility, Québec, Quebec
- Germany (3):
  - Research Facility, Münster, Münster
  - Research Facility, Aachen
  - Research Facility, Hamburg
- United Kingdom (13):
  - Site Facility, Headington, Oxford
  - Research Facility, Solihull, West Midlands
  - Research Facility, Atherstone
  - Research Facility, Coventry
  - Research Facility, Doncaster
  - Research Facility, Headington
  - Research Facility, Herts
  - Research Facility, Leicester
  - Research Facility, Lichfield
  - Research Facility, London
  - Research Facility, Plymouth
  - Research Facility, Salford
  - Research Facility, Warks